CLINICAL TRIAL: NCT00275548
Title: A Prospective, Randomized, Multi-center, Open-label, Comparative Safety and Efficacy Study of Prophylactically Administered Pegylated Interferon Alfa-2a(Pegasys) Plus Ribavirin vs. No Prophylaxis Following Liver Transplantation for Hepatitis C.
Brief Title: Safety and Effectiveness Using Pegasys and Copegus in Recipients of Liver Transplantation With Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Michael R Charlton, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1404-04
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Liver Transplant; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- The Preventative (Prophylaxis) Group: (Other): This group of patients will receive study drugs for the treatment of recurring (or returning) hepatitis C before they actually develop clinical symptoms of hepatitis C.
  Interventions: Drug: Pegasys; Drug: Copegus
- The Observational Group: (Other): This group of patients will receive the study drugs for the treatment of recurring hepatitis C only if they develop the clinical symptoms of hepatitis C infection.
  Interventions: Drug: Pegasys; Drug: Copegus

INTERVENTIONS:
Drug: Pegasys — 135-180 micrograms administered sc once weekly
  Other Names: peginterferon alfa-2a, Ro25-8310)
Drug: Copegus — 400-1200 mg/day for 48 weeks
  Other Names: (ribavirin, Ro20-9963)

SUMMARY:
The study is being done to study the impact of prophylactic administration of antiviral therapy as compared to initiation of antiviral therapy at the time of clinical recurrence of hepatitis C infection in liver transplant recipients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label efficacy and safety study. The study is being done to see whether treatment using Pegasys (pegylated interferon alfa-2a) and Copegus (ribavirin) is safer and more effective in liver transplant recipients when given before hepatitis C infection reappears, or when it is given after clinical symptoms of hepatitis C reinfection appear. The study is also being done in liver transplant recipients to estimate how much hepatitis C is detected over time, how the body affects the study drugs, the safety of the study drugs whether or not the study drugs effect the participants' quality of life, and whether or not the participants feel more or less depressed as a result.

Participants will be put into one of two groups. In the preventive group; participants will receive study drugs for the treatment of recurring (or returning) hepatitis C before developing actual clinical symptoms. The participants in the observational groups will receive study drugs for the treatment of recurring hepatitis C only if they develop the clinical symptoms of hepatitis c infection.

This study will have four parts: a screening phrase, a treatment/observational phrase, follow-up phase and long term safety follow-up phase. Throughout all four stages of the study, participants will have physical exams, medical and surgical history's will be taken, blood and urine tests, eye exam, liver biopsy, chest x-ray and electrocardiogram (ECG). If participants are female, a pregnancy test will also be performed. Participants must also agree not to drink any alcoholic beverages or take any other drugs for hepatitis c infection while taking part in the study. Participants must be able to return for clinic visits at scheduled intervals.

ELIGIBILITY:
Inclusion Criteria:

Positive HCV RNA by PCR at pretransplantation. No biochemical inclusion criteria Male or female patient (>18 yrs) who has undergone liver transplantation because of liver cirrhosis attributed to HCV infection. Patient is a primary, single organ recipient (cadaveric donor). Normal thyroid-stimulating hormone (TSH) Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug. Documentation that female patients of childbearing potential and all male patients are practicing two methods of contraception. For male participants, the following methods are acceptable: 1) vasectomy ANDcondoms with spermicide or 2) vasectomy or condoms with spermicide AND a monogamous relationship with a woman using a single method of contraception. Liver transplant >10 weeks and <26 weeks (6 months) before treatment initiation Patients with a pre-OLT diagnosis of hepatocellular carcinoma (HCC) may be enrolled provided there is no evidence of extrahepatic spread or vascular invasion, and the tumor is solitary and <5 cm or there are up to three tumors <3 cm.

Exclusion Criteria:

Multi-organ or retransplant recipient Patients with HCC who do not meet inclusion criteria or require systemic chemotherapy Recipient of ABO incompatible organ Donor cold ischemia time >20 hrs Anti-HBc positive donor Histological evidence of unresolved rejection Episode of steroid resistant rejection / use of OKT3 Evidence of current Hepatitis B (sAg, cAb, IgM) Seropositivity for HIV infection Serum creatinine >2x upper limit of normal WBC >20,000 x 109/L or ANC <1,500 cells/mm3 Hgb <10g/dL and/or platelets <50,000/mm3 History of autoimmune disease (SLE, scleroderma, rheumatoid arthritis etc.) Uncontrolled seizure disorder Uncontrolled depression or history of suicide attempts/ideation History or evidence of retinopathy Unable or unwilling to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07; Primary Completion 2007-06 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each group who experienced histologically confirmed recurrence of HCV at 120 weeks post randomization. | 96 weeks

SECONDARY OUTCOMES:
The proportion of patients who have non-detectable serum HCV-RNA measured by Quanta Sure plus HCV test and HCV RNA negative by quantitative PCR at week 12, 24, and 48 following initiation of treatment or on observation. | 96 weeks
Virological response rate to antiviral therapy at week 12, week 24, and week 48 of therapy among patients who received antiviral therapy in either study arm. | 96 weeks
Sustained virological response rate: the virological response at the conclusion of the 24 weeks treatment free follow-up period or 72 weeks on observation (for patients who received no treatment). | 96 weeks
The virological response at the conclusion of the 24 weeks treatment-free follow-up period among patients who received antiviral therapy in either arm of the study. | 96 weeks
Patient death or graft failure (as indicated by retransplantation). | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Charlton, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States